CLINICAL TRIAL: NCT05981820
Title: Effect of High Intensity Interval Training and Creatine Intake on Anaerobic Power and Muscle Strength
Brief Title: High Intensity Interval Training, Creatine Intake and Anaerobic Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Dicle Aras, Director, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnkaraUSport
Record Dates: First submitted 2023-04-26; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Creatine; High Intensity Interval Training
Keywords: ergogenic aids; HIIT; creatine; performance
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT group (Experimental): This group will only participate Wingate-based HIIT training.
  In the first three weeks:
  * Warm-up: Warm-up at 70 rpm for 4 minutes, including 2-3 seconds of maximal sprint at 1.30 and 2.30 minutes
  * Wingate-based HIIT: HIIT 4 sets of 12x15 seconds of maximal repetitions with 15 seconds of passive rest between reps in each set
  * Cool-down: 4 minutes of passive rest between sets
  In the last three weeks:
  * Warm-up: Warm-up at 70 rpm for 4 minutes, including 2-3 seconds of maximal sprint at 1.30 and 2.30 minutes
  * Wingate-based HIIT: HIIT 5 sets of 20x15 seconds of maximal repetitions with 15 seconds of passive rest between reps in each set Cool-down: 4 minutes of passive rest between sets
  Interventions: Other: HIIT training
- HIIT + creatine group (Experimental): The HIIT + creatine group will participate the same Wingate-based HIIT training in addition to consume 10 g of creatine supplementation. Participants in this group will use 10 g of creatine monohydrate by dissolved in 200 ml of water. Creatine supplementation will be taken in two doses of five grams, 30 minutes before and after training.
  Interventions: Dietary Supplement: Creatine; Other: HIIT training

INTERVENTIONS:
Dietary Supplement: Creatine — To observe the effects of creatine in the study, 10 g of creatine supplementation was taken only on training days during the study period. Participants used 10 g of creatine monohydrate by dissolved in 200 ml of water. Creatine supplementation was taken in two doses of five grams, 30 minutes before and after training.
  Arms: HIIT + creatine group
Other: HIIT training — In the first three weeks:
  Warm-up: Warm-up at 70 rpm for 4 minutes, including 2-3 seconds of maximal sprint at 1.30 and 2.30 minutes Wingate-based HIIT: HIIT 4 sets of 12x15 seconds of maximal repetitions with 15 seconds of passive rest between reps in each set Cool-down: 4 minutes of passive rest between sets
  In the last three weeks:
  Warm-up: Warm-up at 70 rpm for 4 minutes, including 2-3 seconds of maximal sprint at 1.30 and 2.30 minutes Wingate-based HIIT: HIIT 5 sets of 20x15 seconds of maximal repetitions with 15 seconds of passive rest between reps in each set Cool-down: 4 minutes of passive rest between sets

SUMMARY:
Creatine is an ergogenic aid with positive effects on muscle and performance. The aim of the study was to determine whether there is a difference between the effects of creatine supplementation taken together with Wingate-based HIIT on anaerobic power, leg strength, heart rate variability and body composition. In the study, Wingate-based HIIT program was applied three days a week for six weeks. Anaerobic power (Wingate anaerobic power test), heart rate variability (Polar H10 chest band), leg strength (back and leg dynamometer) and body composition (PlusAvis 333) measurements of the participants were made 1 week before the training program started and the week after the training program ended. Twenty physically active adult men aged 18-30 were voluntarily included for the study. Participants were divided into two groups: Wingate-based HIIT with creatine supplementation (K-HIIT) and Wingate-based HIIT only (HIIT). As a result of the analysis, it was seen that creatine supplementation taken together with wingate-based HIIT had an effect and increased on the anaerobic power parameters, peak power, average power and minimum power values, and leg strength. In addition, it was determined that heart rate variability parameters improved heart rate (HR, beat/min) and low frequency (LF, ms2) values, but did not cause any change in body composition. Comparing and investigating the effects of different HIIT methods on anaerobic power, leg strength, heart rate variability and body composition will increase the generalizability of the study.

DETAILED DESCRIPTION:
Despite the time-efficiency of HIIT in inducing chronic physiological adaptation, it depleted phosphocreatine stores in the muscle and decrease power output. It has been observed that high-intensity exercise performance increases with the increase of intramuscular phosphocreatine. It is thought that with creatine supplementation, the rate of phosphocreatine resynthesis and mitochondrial transfer of ATP to the cytoplasm may increase. This suggests that performing HIIT with creatine supplementation will provide further improvement. Therefore, the purpose of this study to compare the effectiveness of HIIT with creatine supplement compared to HIIT only. We hypothesized that creatine supplementation intake with wingate-based HIIT will positively affect power capacity and performance-related parameters.

The research will be carried out using experimental research design, one of the quantitative research methods, to measure the variables and determine the relationship between dependent and independent variables. Anaerobic power, heart rate variability, leg strength, and body composition measurements of the participants will be made 1 week before the training program started and the week after the training program ended.

The G*power software was utilized in order to determine the appropriate sample size. It has been reported that a minimum of 12 participants, 6 in each group, should be included in the study (alpha value = 0.05, 1-beta value = 0.80, and effect size = 1.6). Measurement of tests and the Wingate-based HIIT program will be conducted in the Performance Laboratory of the Faculty of Sports Sciences of Ankara University. Twenty physically active adult men aged 18-30 years, who had no history of medical and did not use drugs or ergogenic aids, will be recruited voluntarily. The ethics committee approval for the study methodology was obtained from the Ethics Committee of Ankara University Rectorate (Number: E-56786525-050.04.04/378028 Decision Number: 2022/02) and it will be carried out in compliance with the Declaration of Helsinki's principles. Written inform consents which explain the study to the participant and any right and risk will be obtained prior to data collection. Permission for the research to be carried out in the Performance Laboratory of the Faculty of Sport Sciences of Ankara University will be obtained from the Deanery of the Faculty of Sport Sciences of Ankara University. Participants will be divided into two groups as those who will perform Wingate-based HIIT with creatine (C-HIIT) (age: 21,78 ± 1,79 years; height: 179.56 ± 8.26 cm; weight: 76.86 ± 10.66 kg) and those who will perform only Wingate-based HIIT (HIIT) (age: 20.167 ± 0,98 years; height: 172.33 ± 9,88 cm ; weight: 66.53 ± 9.51kg ). Out of twenty potential participants, only 15 participants agreed to participate in the study (HIIT=6, C-HIIT=9) and 5 dropped out because of sport injuries that occured before the study process.

IBM SPSS 24.0 program (SPSS Inc., Chicago, IL, USA) will be used to statistically analyze the data obtained in the study. First of all, the distribution of the data will be evaluated to determine the test used to compare the data as parametric or non-parametric. This normality distribution assessment will be tested with Shapiro Wilk, as both groups had less than 50 participants. Determination of the mean difference in within-group statistics will be performed with Paired Sample t-Test in data with normal distribution and with Wilcoxon test in data where it is not normal. Groups will be expressed as mean ± standard error. American Psychological Association (APA) 6.0 style will be used to report statistical differences. The alpha value will be accepted as 0.05 in all statistical analysis.

This study aimed to determine whether there was a difference in the effects of taking creatine supplementation with Wingate-based HIIT on anaerobic power, leg strength, heart rate variability and body composition.

The limitation of the current research is that the study will be carried out with a single gender. In future studies on the subject, the number of participants can be increased, female participants can be included in the research and it can be examined whether there is a difference between genders and to increase the generalizability of the study, the effects of different HIIT methods on anaerobic power, leg strength, heart rate variability and body composition can be compared by investigating. In addition, the trial period may be extended as longer periods are needed to see clearer changes in HRV.

ELIGIBILITY:
Inclusion Criteria:

* having no health and communication problem
* using no drugs or ergogenic aids
* being physically active adult men aged 18-30 years

Exclusion Criteria:

* using any drugs or ergogenic aids
* having any musculoskeletal problem

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Wingate anaerobic power test | two months
  The Wingate anaerobic power test will be performed using a bicycle ergometer.First, a four-minute warm-up protocol with a bicycle ergometer at 60-80 rpm pedal speed and 50 W workload will be applied. Weights of 7.5% kilograms of their body weight for each participant will be placed on the pan of the bicycle ergometer and anaerobic power testing will be initiated. When they reach the pedal speed to 150 rpm, the test will start. Their maximal effort during 30-seconds will be collected. The Wingate software will be used in which the program set up with the ergometers. Information about the relevant power parameters during the test will be transmitted to the software program on the computer. All power parameters such as both absolute and relative peak power, minimum power, average power etc. will be calculated by the software program automatically.
Leg strength | two months
  Back and leg dynamometer (Takei-Back & Lift, Japan) will be used to measure leg strength. Participants will be placed their feet on the dynamometer stand. The legs will be bent at 15 angles, the body slightly forward, and the back straight. The participants will pull the dynamometer bar, which they grasped with their hands, using only their legs, without changing their current position, until the knees will be extended. Participants will repeat this trial twice, and the best value for each participant will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Dicle Aras, Study Director — Ankara University Faculty of Sport Sciences
Locations (1):
- Ankara University Spor Bilimleri Fakultesi, Gölbaşı, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No